CLINICAL TRIAL: NCT04704076
Title: Preventing Infant Malnutrition With Early Supplementation, Aim 3
Brief Title: Preventing Infant Malnutrition With Early Supplementation
Acronym: PRIMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: International Partnership for Human Development (Unknown); Makerere University (Other); Bill and Melinda Gates Foundation (Other); University of California, Davis (Other); University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-29405
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Underweight; Wasting; Stunting; Breastfeeding; Microbial Colonization
MeSH Terms: conditions — Thinness; Cachexia; Growth Disorders; Breast Feeding; Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early, Small-Volume Supplementation (ESVS) (Experimental): Breastfeeding with up to 59 mL formula daily until 30 days of age, followed by recommendation to breastfeed exclusively through 6 months of age
  Interventions: Other: ESVS
- Exclusive Breastfeeding (Active Comparator): Recommendation to breastfeed exclusively for 6 months without any other food or fluid except vitamins, minerals and medications
  Interventions: Other: Exclusive breastfeeding

INTERVENTIONS:
Other: ESVS — Breastfeeding with up to 59-mL formula daily for the first 30 days, followed by exclusive breastfeeding through 6 months of age
  Arms: Early, Small-Volume Supplementation (ESVS)
Other: Exclusive breastfeeding — Breastfeeding exclusively without any other food or fluid except vitamins, minerals and medications through 6 months of age
  Arms: Exclusive Breastfeeding

SUMMARY:
Background: Worldwide, more than 50 million children under 5 years of age are wasted (weight-for-length/height Z-score (WLZ) <-2) and over 150 million children under 5 are stunted (length/height-for-age Z-score (LAZ) <-2); such wasting and stunting often begin during infancy.1 Optimal nutrition can prevent wasting and stunting. Exclusive breastfeeding (EBF) is widely recommended by community health workers, doctors and nurses and provides optimal nutrition for most infants. However, early growth faltering is common for infants in low and middle income countries (LMIC) and can both increase an infant's risk of early mortality and also lead to deficits in attained height and weight throughout childhood. Thus research is needed to determine the most efficacious strategy to promote healthy early growth in LMIC.

Objective: The proposed study will test the efficacy of early small-volume supplementation (ESVS) for increasing weight-for-age z-score (WAZ) at 1 month of age.

Methodology: The PRIMES pilot (Study 3) will be a randomized clinical trial enrolling infants in Guinea-Bissau and Uganda weighing ≥2000g at birth. Infants weighing 2000-2499g at <6 hours of age (n=144; 72 per site) will be randomized on enrollment to one of two groups: 1) Early Small-Volume Supplementation (ESVS intervention group), which consists of up to 59 mL formula administered daily after breastfeeding through 30 days of age followed by EBF through 6 months of age; or 2) frequent exclusive breastfeeding without any food or fluid other than vitamins, minerals and medications (control) through 6 months of age. Infants weighing 2500-3300g at <6 hours of age will be weighed again at 4 days of age; those weighing <2600g at 4 days of age (n=180; 90 per site) will be randomized to the same intervention and control groups. Weight will be measured on all enrolled babies at birth on Day 1 and at 4, 14, 30, 60 and 180 days of age and additional measures including height, MUAC, skinfolds, and hemoglobin will be assessed at other time points. The study's primary outcome will be WAZ at 1 month of age. Secondary outcomes will include WLZ at 1 month of age; WAZ, WLZ and LAZ through 6 months of age; breastfeeding duration and infant intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Infant < 6 hours old
* Infant birth weight 2000-2885g
* Mother intends to breastfeed
* Mother with negative HIV test
* Mother lives in study catchment area and anticipates availability for all study visits
* Mother ≥18 years old

Exclusion Criteria:

* Twins and other multiples
* Infant with known major congenital anomalies including orofacial clefts, neural tube defects or congenital heart defects
* Infant with WHO newborn and respiratory danger signs present:

  * Not feeding well
  * Convulsions
  * Very fast breathing ≥60 breaths/minute
  * Severe chest indrawing
  * No spontaneous movement
  * Lethargic or unconscious
  * Raised temperature > 37.5 degrees Celsius
  * Hypothermia <35.5 degrees Celsius
  * Any jaundice in first 24 hours of life or yellow palms or soles at any age
  * Head nodding, nasal flaring or grunting
* Maternal psychiatric or psychosocial barrier to enrollment:

  * Contraindication to breastfeeding at each site as determined by a site's national or sub-national health authorities
  * Mothers unable or unwilling to complete all aspects of the protocol Infant enrolled in another study
  * Mother has had another infant enrolled in PRIMES

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Weight-for-age z-score (WAZ) at 30 days of age | 30 days of age
  WAZ calculated according to WHO Child Growth Standards

SECONDARY OUTCOMES:
Weight-for-length z-score (WLZ) at 30 days of age | 30 days of age
  WLZ calculated according to WHO Child Growth Standards
Weight-for-length z-score (WLZ) at 180 days of age | 180 days of age
  WLZ calculated according to WHO Child Growth Standards
Weight-for-length z-score (WLZ) at 365 days of age | 365 days of age
  WLZ calculated according to WHO Child Growth Standards
Weight-for-age z-score (WLZ) at 180 days of age | 180 days of age
  WAZ calculated according to WHO Child Growth Standards
Weight-for-age z-score (WLZ) at 365 days of age | 365 days of age
  WAZ calculated according to WHO Child Growth Standards
Length-for-age z-score (LAZ) at 180 days of age | 180 days of age
  LAZ calculated according to WHO Child Growth Standards
Length-for-age z-score (LAZ) at 365 days of age | 365 days of age
  LAZ calculated according to WHO Child Growth Standards
Whether or not breastfeeding continues at 180 days of age | 180 days of age
  Continuation of breastfeeding
Abundance of B.infantis in intestinal microbiota | 30 days of age
  Microbiota will be collected in DNA/RNA Shield Fecal Collection Tube containers (Zymo Research, Irvine, CA) and analyzed using 16S rRNA gene profiling
Abundance of B.infantis in intestinal microbiota | 180 days of age
  Microbiota will be collected in DNA/RNA Shield Fecal Collection Tube containers (Zymo Research, Irvine, CA) and analyzed using 16S rRNA gene profiling
Neurodevelopment | 180 days of age
  Bayley Scales of Infant and Toddler Development, 3rd Edition
Neurodevelopment | 365 days of age
  Bayley Scales of Infant and Toddler Development, 3rd Edition
Brain volume | 90 days of age
  Low-field MRI
Brain volume | 180 days of age
  Low-field MRI
Brain volume | 365 days of age
  Low-field MRI
White matter volume | 365 days of age
  Conventional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flaherman, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- International Partnership for Human Development, Bissau, Guinea-Bissau
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ginsburg AS, Braima de Sa A, Nankabirwa V, Co R, Murungi J, Kim MO, Brim R, Namiiro F, Namugga O, Hartigan-O'Connor DJ, Roberts SB, Flaherman V. Randomized controlled trial of early, small-volume formula supplementation among newborns: A study protocol. PLoS One. 2022 Feb 4;17(2):e0263129. doi: 10.1371/journal.pone.0263129. eCollection 2022. PMID 35120150